CLINICAL TRIAL: NCT03822416
Title: Treating Tobacco Dependence in Smokers With Severe Mental Illness
Brief Title: Treating Smokers With Mental Illness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Hennepin County Medical Center, Minneapolis (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPH-2018-26854
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Smoking Cessation; Cigarette Smoking; Schizophrenia; Psychotic Disorders; Major Depressive Disorder; Bipolar Disorder I; Bipolar II Disorder; Mental Illness
Keywords: mental illness; tobacco treatment
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking; Schizophrenia; Psychotic Disorders; Depressive Disorder, Major; Bipolar Disorder; Mental Disorders | interventions — Tobacco Use Cessation Devices; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not be made aware of the participant's study status, although it may become obvious during the assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group will receive counseling and nicotine replacement therapy including the nicotine patch and/or nicotine lozenges.
  Interventions: Drug: Nicotine patch; Drug: Nicotine lozenge; Behavioral: Therapy; Other: Information
- Control (Other): Control group will receive information about mental illness and smoking cessation and a listing of community resources available for assistance with smoking cessation.
  Interventions: Other: Information

INTERVENTIONS:
Drug: Nicotine patch — Nicotine patch (dose based on number of cigarettes per day) (4-week, 8-week, or 12-week supply) depending on participant preference and how much they are smoking based on FDA guidelines for use
  Arms: Intervention
Drug: Nicotine lozenge — Nicotine lozenge (2 or 4 mg if less or greater than 30 minutes to first cigarette in the morning respectively) (4-week, 8-week, or 12-week supply) depending on participant preference and how much they are smoking based on FDA guidelines for use
  Arms: Intervention
Behavioral: Therapy — In-person meeting at baseline, 6 phone counseling sessions with participants over 8 weeks after initial in-person meeting, possible additional phone counseling (3 phone calls) from 8 weeks to 6 months after initial in-person meeting, and possible text messages when agreed to by participants during the 8 week to 6 month phase
  Arms: Intervention
Other: Information — Information about smoking and mental illness and referrals to both the QUITPLAN helpline and additional resources in the community

SUMMARY:
This is a smoking cessation study that will enroll smokers who have been diagnosed with a severe mental illness. The study will use a combination of intensive tobacco treatment counseling and nicotine replacement therapy to assist smokers in cutting back on and quitting smoking over the course of six months.

DETAILED DESCRIPTION:
At the baseline measurement visit, participants will be asked to complete a survey and an interview. They will be randomly assigned to either the intervention or control group. Both groups will receive a smoking cessation manual and list of resources. The intervention group will also receive smoking cessation counseling and nicotine replacement therapy. Both groups will be seen for in-person assessments again at 8 weeks and 6 months post baseline.

ELIGIBILITY:
Inclusion Criteria:

* have a severe mental illness diagnosis
* be a daily smoker
* be willing to reduce the number of cigarettes smoked per day leading to a quit attempt
* want to try to quit smoking
* be willing to use nicotine replacement therapy
* be able to communicate in English

Exclusion Criteria:

* anyone who has had an active psychotic episode or been hospitalized due to suicidal ideation in the last six months
* pregnancy
* taking Chantix or Clozapine
* having a terminal illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Lando, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Busch AM, Nederhoff DM, Dunsiger SI, Japuntich SJ, Chrastek M, Adkins-Hempel M, Rinehart LM, Lando H. Chronic care treatment for smoking cessation in patients with serious mental illness: a pilot randomized trial. BMC Psychiatry. 2021 Feb 17;21(1):104. doi: 10.1186/s12888-021-03113-5. PMID 33593332

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 19 | 19
Completed | 18 | 18
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 1 | 0 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 11 | 7 | 18
  Other | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 8 | 10 | 18
  More than one race | 1 | 6 | 7
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: 7-Day Point Prevalence Abstinence
Description: To determine the number of patients in the intervention and control conditions who achieve 7-day point prevalence abstinence at 8 weeks and 6 months after enrollment.
Time Frame: 8 weeks and 6 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 19
Participants
  8 Weeks | 5 | 3
  6 Months | 4 | 5

2. Secondary Outcome: Quit Attempts
Description: To determine the number of patients in the intervention and control condition who achieve self-reported minimum 24 hour quit attempts.
Time Frame: 8 weeks and 6 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 19
Participants
  8 Weeks | 13 | 7
  6 Months | 18 | 10

3. Secondary Outcome: Smoking Reduction
Description: To determine the mean reduction in cigarettes per day in the intervention and control conditions.
Time Frame: 8 weeks and 6 months post baseline
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 19
cigarettes per day
  8 Weeks | 5.6 (7.04) | 11.59 (4.15)
  6 Months | 4.84 (4.56) | 8.03 (3.23)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 1/19 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=19) | Control (N=19)
increased coughing following smoking cessation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT03822416/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT03822416/ICF_001.pdf